CLINICAL TRIAL: NCT02349841
Title: A Phase 2 Trial to Evaluate the Early Bactericidal Activity, Safety and Tolerability of Meropenem, Administered Intravenously, Plus Amoxycillin/CA and Faropenem, Administered Orally, Plus Amoxycillin/CA in Adult Patients With Newly Diagnosed, Smear-positive Pulmonary Tuberculosis.
Brief Title: Phase 2 Trial to Evaluate the Early Bactericidal Activity, Safety and Tolerability of Meropenem Plus Amoxycillin/CA and Faropenem Plus Amoxycillin/CA in Adult Patients With Newly Diagnosed Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TASK Applied Science (Other)
Collaborators: Eduardo Mondlane University (Other); GlaxoSmithKline (Industry); Barcelona Centre for International Health Research (Other); Research Center Borstel (Other)
Responsible Party: Principal Investigator, Andreas Henri Diacon, Professor Andreas H Diacon, TASK Applied Science
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASK-001
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Meropenem; fropenem; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meropenem;amoxycillin/clavulanic acid (Experimental): Meropenem 2g will be administered intravenously 8-hourly; plus amoxycillin/CA 500mg/125mg will be administered orally 8-hourly for 14 days
  Interventions: Drug: Meropenem; Drug: Amoxycillin/clavulanic acid
- Faropenem; amoxycillin/CA (Experimental): Faropenem 600mg will be administered orally 8-hourly; plus amoxycillin/CA 500mg/125mg will be administered orally 8-hourly for 14 days
  Interventions: Drug: Faropenem; Drug: Amoxycillin/clavulanic acid
- Rifafour e-275 (Active Comparator): Rifafour e-275 will be administered orally once daily for 14 days as per South African National TB Treatment Guidelines
  Interventions: Drug: Rifafour e275

INTERVENTIONS:
Drug: Meropenem — To administer 2g daily 8 hourly for 14 days
  Arms: Meropenem;amoxycillin/clavulanic acid
Drug: Faropenem — To adminster 600mg 8 hourly daily for 14 days
  Arms: Faropenem; amoxycillin/CA
Drug: Amoxycillin/clavulanic acid — To administer 625mg 8 hourly daily for 14 days together with the faropenem and meropenem
  Arms: Faropenem; amoxycillin/CA; Meropenem;amoxycillin/clavulanic acid
Drug: Rifafour e275 — To be taken as per the National TB treatment programme for 14 days
  Arms: Rifafour e-275

SUMMARY:
To evaluate the early bactericidal activity (EBA), safety, tolerability and pharmacokinetics of meropenem administered intravenously three times a day, plus amoxycillin/CA administered orally three times a day; and of faropenem administered orally three times a day, plus amoxycillin/CA administered orally three times a day; for 14 consecutive days, in adult participants with newly diagnosed, smear positive pulmonary tuberculosis, in order to help establish proof-of-concept for carbapenem antibiotics as antituberculosis agents and to select the appropriate agent and route of administration for later stage clinical development.

DETAILED DESCRIPTION:
A single-centre, open-label clinical trial including a total of 45 male or female participants (2 groups of 15 participants receiving an IMP and 1 group of 15 participants receiving Rifafour e-275), aged between 18 and 65 years (inclusive), with newly diagnosed, smear-positive, pulmonary tuberculosis will be enrolled into this trial.

Treatment will be administered for 14 consecutive days in the following dosing schemes:

1. Meropenem 2g intravenously 8-hourly; plus amoxycillin/CA 500mg/125mg orally 8- hourly on days 1-14.
2. Faropenem 600mg orally 8-hourly; plus amoxycillin/CA 500mg/125mg orally 8-hourly on days 1-14.
3. The third arm will receive standard first line TB treatment as per the South African TB guidelines (Rifafour e-275) and is included as a control for the EBA quantitative mycobacteriology and to evaluate whether HRZE gives similar EBA results to that demonstrated in prior studies with this combination. The mycobacteriology laboratory will remain blinded until closure of the EBA results.

Participants will be admitted to the in hospital facility for a period of up to 24 days. During this period they will await their screening results after which they will receive 14 day of IMP. on day 14 intensive PK sampling will be done. They will be discharged on day 15 to the clinic where they will continue on the national TB programme treatment regime. Participants will return to the clinical trial site 14 days after receipt of their last study drug. for a safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures including HIV testing.
2. Male or female, aged between 18 and 65 years, inclusive.
3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Newly diagnosed, previously untreated, pulmonary TB.
5. A chest X-ray picture which in the opinion of the Investigator is consistent with TB.
6. Sputum positive GeneXpert or TB smear from TB clinic or site of initial diagnosis.
7. Sputum positive on direct microscopy for acid-fast bacilli on at least one sputum sample at the trial appointed laboratory(at least 1+ on the IUATLD/WHO scale).
8. Ability to produce an adequate volume of sputum as estimated from a spot assessment (estimated 10 ml or more overnight production).
9. Be of non-childbearing potential or using effective methods of birth control, as defined below:

Non-childbearing potential:

1. Participant - not heterosexually active or practice sexual abstinence; or
2. Female participant/sexual partner - bilateral oophorectomy, bilateral tubal ligation and/or hysterectomy or has been postmenopausal with a history of no menses for at least 12 consecutive months; or
3. Male participant/sexual partner - vasectomised or has had a bilateral orchidectomy minimally three month prior to screening;

Effective birth control methods:

1. Double barrier method which can include a male condom, diaphragm, cervical cap, or female condom; or
2. Barrier method combined with hormone-based contraceptives or an intra-uterine device for the female partner; and are willing to continue practicing birth control methods throughout participation in the study until Visit 19 (day 28). (Note: hormone-based contraception alone may not be reliable when taking IMP; therefore, hormone-based contraceptives alone cannot be used by female participants to prevent pregnancy).

Exclusion Criteria Medical History

1. Evidence of clinically significant (as judged by the investigator), metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied) including malaria.
2. Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
3. A history of previous TB less than 5 years ago.
4. Clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
5. History of allergy to any of the trial IMP/s or related substances i.e. β-lactams and penicillin, as confirmed by the clinical judgement of the Investigator.
6. Isoniazid-resistant and/or rifampicin-resistant bacteria detected with a sputum specimen collected within the pre-treatment period and tested at the study laboratory.
7. Known or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the participant.
8. For HIV infected participants:

   1. having a CD4+ count <350 cells/µL;
   2. or having received antiretroviral therapy medication within the last 90 days;
   3. or having received oral or intravenous antifungal medication within the last 90 days;
   4. or with an AIDS-defining opportunistic infection or malignancies (except pulmonary TB).
9. Having participated in other clinical studies with investigational agents within 8 weeks prior to trial start.
10. Female participant who is pregnant, breast-feeding, or planning to conceive a child within the anticipated period of participating in the trial. Male participant planning to conceive a child within the anticipated period of participating in the trial.
11. Diabetes mellitus requiring insulin.

    Specific Treatments
12. Treatment received with any drug active against MTB within the 3 months prior to Visit 1 (including but not limited to isoniazid, ethambutol, amikacin, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides, metronidazole).
13. Participants receiving sodium valproate, furosemide, imipenem or probenecid.
14. Any diseases or conditions in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to allergy to any TB drug, their component or to the IMP.

    Laboratory Abnormalities
15. Participants with the following toxicities at screening as defined by the enhanced CTCEA toxicity table

    1. creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]);
    2. hemoglobin grade 4 (<6.5 g/dL);
    3. platelets grade 2 or greater (under 50x109 cells/L);
    4. serum potassium grade 2 or greater (<3.0 mEq/L);
    5. aspartate aminotransferase (AST) grade 3 (≥3.0 x ULN) to be excluded;
    6. alanine aminotransferase (ALT) grade 3 (≥3.0 x ULN) to be excluded;
    7. APTT grade 3
    8. INR grade 3
    9. Total white cell count grade 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint (The EBA CFU(0-14) as determined by the rate of change in logCFU per ml sputum) | 14 days
  The EBA CFU(0-14) as determined by the rate of change in logCFU per ml sputum over the period Day 0 to Day 14 which will be described with at most 3 parameters from a linear, bi-linear or non-linear regression of logCFU on time

SECONDARY OUTCOMES:
Efficacy (The EBA CFU(0-2) and EBA CFU(2-14) as determined by the rate of change of logCFU in sputum) | 14 days
  The EBA CFU(0-2) and EBA CFU(2-14) as determined by the rate of change of logCFU in sputum over the period Day 0 to Day 2 and Day 2 to Day 14, which will be described with at most 3 parameters from an appropriate function of logCFU on time.
  The EBA TTP(0-2), EBA TTP(0-14), and EBA TTP(2-14) in the Mycobacterial Growth Indicator Tube (BactecTM MGITTM 960) system as determined by the rate of change in TTP in sputum over the periods Day 0 to Day 2, Day 0 to Day 14, and will be described with at most 3 parameters from an appropriate function of TTP on time.
Safety and Tolerability (Incidence of treatment emergent adverse events (TEAEs) | 28 days
  will be presented by severity, IMP relatedness, seriousness, leading to early withdrawal and leading to death
Pharmacokinetics (The maximum observed plasma concentration (Cmax), time to reach Cmax (Tmax), the minimum observed plasma concentration (Cmin) | 14 days
  The maximum observed plasma concentration (Cmax), time to reach Cmax (Tmax), the minimum observed plasma concentration (Cmin) 24 hours following the intake if the first daily dosing on day 14, area under the plasma concentration time (t) curve from zero to 24 hours (AUC(0-24)) will be estimated for the following, on Day 14
Pharmacokinetics - Pharmacodynamics (descriptive analyses, and no inferential tests will be carried out, of EBA CFU(0-14), EBA CFU(0-2), and EBA CFU(2-14) vs. AUC(0-24) • Time over Minimum inhibitory concentrations (TMIC) (for meropenem; faropenem) | 14 days
  The EBA CFU(0-14), EBA CFU(0-2), and EBA CFU(2-14) vs. the following PK variables will be presented for meropenem and faropenem:
  * Cmax
  * AUC(0-24)
  * Time over Minimum inhibitory concentrations (TMIC) (for meropenem; faropenem)
  * These data will be presented as descriptive analyses, and no inferential tests will be carried out.

CONTACTS AND LOCATIONS:
Locations (1):
- TASK Foundation NPC, Cape Town, Western Cape, South Africa